CLINICAL TRIAL: NCT02125747
Title: Effectiveness of Respiratory Therapy in Acute Exacerbations of Chronic Obstructive Pulmonary Disease
Brief Title: Respiratory Therapy in COPD Exacerbations
Acronym: TRESEPOCAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Esther Marco Navarro, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSM/RHB/CR/05
Record Dates: First submitted 2014-04-23; First posted 2014-04-29 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2015-04

CONDITIONS: Obstructive Chronic Bronchitis With Acute Exacerbation
Keywords: Respiratory muscle training; high-intensity training
MeSH Terms: interventions — Respiratory Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Respiratory Therapy (Other): Patients with acute exacerbation of chronic obstructive pulmonary disease. Patients received conventional treatment.
  Interventions: Other: No Respiratory Therapy
- Respiratory therapy (Experimental): Patients with acute exacerbation of chronic obstructive pulmonary disease. Patients received conventional treatment and Respiratory Therapy
  Interventions: Other: Respiratory Therapy

INTERVENTIONS:
Other: No Respiratory Therapy — Patients received conventional treatment.
  Arms: No Respiratory Therapy
Other: Respiratory Therapy — Respiratory Therapy consists of postural drainage, positive expiratory pressure (PEP) and vibropercussion (it is a postural drainage method, which uses chest clapping with a flexible wrist and cupped hands or a mechanical vibrator to loosen and mobilize retained secretions that can then be expectorated or drained). Postural drainage is an airways clearance technique in which patient's body is positioned so that the trachea is inclined downward and below the affected chest area.
  The PEP consists of expiratory cycles through a system generating a positive pressure of 10-20 cc (cubic centimeter) water. Vibropercussion is applied by the use of a mechanical system following rib movement during expiration to enhance clearance of secretions.
  Intervention group received 30-minute-sessions twice a day, 7 days per week, during hospitalization period.
  Arms: Respiratory therapy

SUMMARY:
The purpose of this study is to determine effectiveness, feasibility and safety/tolerance of Respiratory Therapy in hospitalized patients with acute exacerbations of chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Acute exacerbation of chronic obstructive pulmonary disease (AE-COPD) is defined as an event in the natural course of the disease characterized by a change in the patient's usual symptoms (dyspnea, cough and/or sputum) that may not be explained by the daily variations and requires a change in regular medication.

Because AE-COPD result in impairment of both pulmonary and respiratory muscle functions, as well as an increasing impact on costs, priority should be given to interventions to slow the progression of the disease, prevention of exacerbations and reduce the risk of comorbidity.

Chest physiotherapy is often used in hospitalized patients with AE-COPD with the aim of favoring the removal of secretions and thus to improve the ventilation perfusion (V/Q), and therefore the function lung. The limited scientific evidence has determined that their use is controversial and not routinely recommended in clinical practice guidelines. Current clinical guidelines in the treatment of COPD are unable to rule on the application of respiratory therapy during exacerbations, since there is little scientific evidence of its benefits in the short and long term.

ELIGIBILITY:
Hospitalized patients with acute exacerbation of COPD.

Inclusion Criteria:

* age over 18 years,
* hospitalized patients and
* acute exacerbation of COPD.

Exclusion Criteria:

* Previous history of any chronic respiratory disease and
* not to have performed any kind of general or respiratory training in the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-12; Primary Completion 2012-05 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strength | Participants will be followed for the duration of hospital stay, an expected average of 10 days
  Respiratory muscle strength is assessed through maximal inspiratory pressures (MIP) and maximal expiratory pressures (MEP) using a pressure transducer connected to a digital register system. The MIP is measured at mouth during a maximum effort from residual volume against occluded airway. To determine the MEP, patients performed a maximum expiratory effort from total lung capacity in the face of the occluded airway.

SECONDARY OUTCOMES:
Measure of safety and tolerability | Participants will be followed for the duration of hospital stay, an expected average of 10 days
  Presence of complications and patients' satisfaction
Adverse events as a measure of safety and tolerability | One year after hospital discharge
  Monitoring of health status and possible complications one year after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Orozco-Levi, MD, PhD, Study Director — Biomedical Research Network for Respiratory Diseases (CIBERES), ISCIII, Ministerio de Ciencia y Tecnología, Spain; Respiratory Department, Hospital del Mar, Spain; Respiratory Department, Centro de Investigaciones, Fundación Cardiovascular de Colombia
Locations (1):
- Departments of Respiratory Medicine and Rehabilitation. Parc de Salut Mar, Hospital del Mar, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Jones AP, Rowe BH. Bronchopulmonary hygiene physical therapy for chronic obstructive pulmonary disease and bronchiectasis. Cochrane Database Syst Rev. 2000;(2):CD000045. doi: 10.1002/14651858.CD000045. PMID 10796474
- [Background] Sivasothy P, Brown L, Smith IE, Shneerson JM. Effect of manually assisted cough and mechanical insufflation on cough flow of normal subjects, patients with chronic obstructive pulmonary disease (COPD), and patients with respiratory muscle weakness. Thorax. 2001 Jun;56(6):438-44. doi: 10.1136/thorax.56.6.438. PMID 11359958
- [Background] Gulsvik A. The global burden and impact of chronic obstructive pulmonary disease worldwide. Monaldi Arch Chest Dis. 2001 Jun;56(3):261-4. PMID 11665507
- [Background] Elkins MR, Jones A, van der Schans C. Positive expiratory pressure physiotherapy for airway clearance in people with cystic fibrosis. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD003147. doi: 10.1002/14651858.CD003147.pub3. PMID 16625571
- [Background] Standards for the diagnosis and care of patients with chronic obstructive pulmonary disease. American Thoracic Society. Am J Respir Crit Care Med. 1995 Nov;152(5 Pt 2):S77-121. No abstract available. PMID 7582322
- [Background] Puhan MA, Scharplatz M, Troosters T, Steurer J. Respiratory rehabilitation after acute exacerbation of COPD may reduce risk for readmission and mortality -- a systematic review. Respir Res. 2005 Jun 8;6(1):54. doi: 10.1186/1465-9921-6-54. PMID 15943867
- [Background] Olseni L, Midgren B, Hornblad Y, Wollmer P. Chest physiotherapy in chronic obstructive pulmonary disease: forced expiratory technique combined with either postural drainage or positive expiratory pressure breathing. Respir Med. 1994 Jul;88(6):435-40. doi: 10.1016/s0954-6111(05)80046-0. PMID 7938794
- [Background] Hill K, Patman S, Brooks D. Effect of airway clearance techniques in patients experiencing an acute exacerbation of chronic obstructive pulmonary disease: a systematic review. Chron Respir Dis. 2010;7(1):9-17. doi: 10.1177/1479972309348659. Epub 2009 Oct 9. PMID 19819912
- [Background] Mohsenifar Z, Rosenberg N, Goldberg HS, Koerner SK. Mechanical vibration and conventional chest physiotherapy in outpatients with stable chronic obstructive lung disease. Chest. 1985 Apr;87(4):483-5. doi: 10.1378/chest.87.4.483. PMID 3884288
- [Background] Miravitlles M, Ferrer M, Pont A, Zalacain R, Alvarez-Sala JL, Masa F, Verea H, Murio C, Ros F, Vidal R; IMPAC Study Group. Effect of exacerbations on quality of life in patients with chronic obstructive pulmonary disease: a 2 year follow up study. Thorax. 2004 May;59(5):387-95. doi: 10.1136/thx.2003.008730. PMID 15115864
- [Background] Newton DA, Stephenson A. Effect of physiotherapy on pulmonary function. A laboratory study. Lancet. 1978 Jul 29;2(8083):228-9. doi: 10.1016/s0140-6736(78)91742-7. PMID 79027
- [Background] Garrod R, Lasserson T. Role of physiotherapy in the management of chronic lung diseases: an overview of systematic reviews. Respir Med. 2007 Dec;101(12):2429-36. doi: 10.1016/j.rmed.2007.06.007. Epub 2007 Sep 17. PMID 17870457
- [Background] Tang CY, Taylor NF, Blackstock FC. Chest physiotherapy for patients admitted to hospital with an acute exacerbation of chronic obstructive pulmonary disease (COPD): a systematic review. Physiotherapy. 2010 Mar;96(1):1-13. doi: 10.1016/j.physio.2009.06.008. Epub 2009 Sep 22. PMID 20113757
- [Background] Lange P, Nyboe J, Appleyard M, Jensen G, Schnohr P. Relation of ventilatory impairment and of chronic mucus hypersecretion to mortality from obstructive lung disease and from all causes. Thorax. 1990 Aug;45(8):579-85. doi: 10.1136/thx.45.8.579. PMID 2402719
- [Background] Opdekamp C, Sergysels R. [Respiratory physiotherapy in lung diseases]. Rev Med Brux. 2003 Sep;24(4):A231-5. French. PMID 14606285
- [Background] Wolkove N, Kamel H, Rotaple M, Baltzan MA Jr. Use of a mucus clearance device enhances the bronchodilator response in patients with stable COPD. Chest. 2002 Mar;121(3):702-7. doi: 10.1378/chest.121.3.702. PMID 11888949
- [Background] Ides K, Vissers D, De Backer L, Leemans G, De Backer W. Airway clearance in COPD: need for a breath of fresh air? A systematic review. COPD. 2011 Jun;8(3):196-205. doi: 10.3109/15412555.2011.560582. Epub 2011 Apr 22. PMID 21513439
- [Background] van der Schans CP. Conventional chest physical therapy for obstructive lung disease. Respir Care. 2007 Sep;52(9):1198-206; discussion 1206-9. PMID 17716386
- [Background] Osadnik CR, McDonald CF, Jones AP, Holland AE. Airway clearance techniques for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD008328. doi: 10.1002/14651858.CD008328.pub2. PMID 22419331